CLINICAL TRIAL: NCT01614639
Title: A Physiological fMRI Study of Acupuncture and Perceptions of Pain in Chronic Low Back Pain Patients.
Brief Title: Brain Imaging Study of Acupuncture in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Robert Edwards, Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2011P000748; P01AT006663-01 (NIH)
Record Dates: First submitted 2012-05-23; First posted 2012-06-08 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Low Back Pain; Back Pain Lower Back Chronic; Low Back Pain, Recurrent
Keywords: Acupuncture; fMRI; CLBP; Pain; Low Back Pain; Back Pain
MeSH Terms: conditions — Low Back Pain; Pain; Back Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional Acupuncture (Experimental): Traditional Acupuncture given at 2 visits.
  Interventions: Procedure: Acupuncture
- Electroacupuncture (Experimental): Electro-acupuncture given at 2 visits.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — A licensed acupuncturist will perform acupuncture for two 30 minute sessions.

SUMMARY:
We are doing this research study to learn about how acupuncture treatment works. This study is being done to look at changes in the brain, NOT to treat pain. We want to learn about brain activity during acupuncture. We will look at brain activity when a heating device touches the skin of a subject before and after the subject has acupuncture, to see what changes.

ELIGIBILITY:
Inclusion Criteria:

* Meet the Classification Criteria of chronic LBP (having low back pain for more than 6 months), as determined by the referring physician
* At least 4/10 clinical pain on the 10-point LBP intensity scale on average during the past two weeks prior to enrollment
* At least a 10th grade English-reading level; English can be a second language provided that the patients feel they understand all the questions used in the assessment measures
* Must have had a prior evaluation of their low back pain by a health care provider, which may include radiographic studies. Documentation of this evaluation will be obtained from the subject's medical record

Exclusion Criteria:

* Specific causes of back pain (e.g., cancer, fractures, spinal stenosis, infections)
* Radicular pain extending below the knee
* Complicated back problems (e.g., prior back surgery, medicolegal issues)
* Possible contraindications for acupuncture (e.g., coagulation disorders, cardiac pacemakers, pregnancy, seizure disorder), and conditions that might confound treatment effects or interpretation of results (e.g., severe fibromyalgia, rheumatoid arthritis)
* Conditions making study participation difficult (e.g., paralysis, psychoses, or other severe psychological problems as per the judgment of a study investigator and/or a T score > 60 on the psychological measures assessed during Session 1)
* Prior acupuncture treatment for back pain; 1 year minimum wait for any condition other condition.
* Active substance abuse disorder in the past two years, as determined by subject self-report.
* The intent to undergo surgery during the time of involvement in the study.
* History of cardiac, respiratory, or nervous system disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for adverse outcome. For example: asthma or claustrophobia.
* Presence of any contraindications to MRI scanning. For example: cardiac pacemaker, metal implants, fear of closed spaces, pregnancy.
* Unresolved legal/disability/workers compensation claims in connection with low back.
* Instability of pain ratings in Session 2 or Session 3.
* Use of more than 60 mg prescription opioids or steroids for pain.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Brain changes to acupuncture | 3 visits
  The effects of pain on the brain

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Edwards, Ph.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- MGH - Martinos Center, Charlestown, Massachusetts, United States